CLINICAL TRIAL: NCT02291731
Title: Topical Autologous Serum Eye Drops Combined With Silicone Hydrogen Lenses for theTreatment of Corneal Epithelial Defects
Brief Title: Autologous Serum Eye Drops With Contact Lenses for Corneal Epithelial Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: E-DA Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: EMRP37103N
Record Dates: First submitted 2014-11-07; First posted 2014-11-14 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Corneal Diseases
Keywords: Autologous serum eye drops; Silicone-hydrogel contact lens; Persistent epithelial defects; Corneal epithelial defects
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Continuous use of autologous serum (Experimental): with continuous use of topical autologous serum for an additional 2 weeks after total re-epithelialization.
  Interventions: Drug: Continuous use of topical autologous serum

INTERVENTIONS:
Drug: Continuous use of topical autologous serum — Silicone-hydrogel SCLs combined with 20% (v/v) autologous serum eye drops were used until complete re-epithelialization. SCLs were removed after total re-epithelialization and patients were subsequently randomized divided into two groups: (1) with and (2) without continuous use of topical autologous serum for an additional 2 weeks after SCLs removal.
  Other Names: autologous serum eye drops

SUMMARY:
To evaluate the clinical effect of combination of topical 20% (v/v) autologous serum eye drops and a silicone-hydrogel contact lens (CLs) in the treatment of recalcitrant persistent epithelial defects (PEDs) and the recurrence rate of epithelial breakdown with or without continued use of autologous serum eye drops.

DETAILED DESCRIPTION:
Dealing with persistent epithelial defects (PEDs) of the cornea is a challenge for ophthalmologists, and surgical intervention is occasionally indicated for the management of recalcitrant cases that are unresponsive to medical therapy. Bandage contact lenses (BCLs), especially silicone-hydrogel CLs with high oxygen permeability and transmissibility, are useful for treating PEDs. Over the past several years, autologous serum eye drops (ASEs) are gaining popular and widespread acceptance as adjuvant therapy for various ocular surface disorders, including PEDs recalcitrant to standard medical therapies.The combination of BCLs and ASEs for PEDs treatment have also been reported with satisfactory results in a few small series' of PED patients. In this study, we will conduct a prospective interventional study to investigate the therapeutic effects of the combination of topical 20% ASEs and silicone-hydrogel CLs for recalcitrant PEDs, as well as to compare the recurrence of epithelial breakdown with or without continuous usage of autologous serum eye drops after CL removal. Patients with PEDs for more than 4 weeks without improvement despite previous conventional treatment were treated. Silicone-hydrogel SCLs combined with 20% (v/v) autologous serum eye drops were used until complete re-epithelialization. SCLs were removed after total re-epithelialization and patients were subsequently randomized divided into two groups: (1) with and (2) without continuous use of topical autologous serum for an additional 2 weeks. PED healing rate and epithelial defect recurrence during a 3-month follow-up were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PEDs for more than 1-month following conventional treatment, visiting E-Da Hospital, Kaohsiung, Taiwan.

Exclusion Criteria:

* Patients had dry eye syndrome with a Schirmer test (<10 mm in 5 minutes) or lid abnormalities.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
epithelial defect healing rate | 2-week

SECONDARY OUTCOMES:
epithelial defect recurrence rate | 3-month

CONTACTS AND LOCATIONS:
Overall Officials: Yan-Ming Chen, M.D., Study Chair — Department of Ophthalmology, E-Da Hospital, I-Shou University, Kaohsiung, Taiwan
Locations (1):
- E-DA hospital, Kaohsiung City, Taiwan